CLINICAL TRIAL: NCT06516445
Title: A Clinical Study of Short Course Radiotherapy (SCRT) Followed by Camrelizumab Combined With Fluzoparib and Chemotherapy as Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Brief Title: SCRT Followed by Camrelizumab Combined With Fluzoparib and Chemotherapy as Neoadjuvant Therapy for LARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-CRC-II-007
Record Dates: First submitted 2024-07-09; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — camrelizumab; fluzoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCRT followed by camrelizumab combined with fluzoparib and chemotherapy (Experimental)
  Interventions: Radiation: SCRT; Drug: Camrelizumab; Drug: Fluzoparib; Drug: CAPEOX

INTERVENTIONS:
Radiation: SCRT — 5×5Gy，5Gy/d，QD，D1-D5
Drug: Camrelizumab — 200mg, D1, ivgtt, Q3W, C1-4
Drug: Fluzoparib — 100mg, BID, PO, Q3W, C1-4
Drug: CAPEOX — Capecitabine: 1000 mg/m2, BID, PO，D1-14, Q3W, C1-C4； Oxaliplatin: 130mg/m2, D1, ivgtt, 0-2h，Q3W，C1-4

SUMMARY:
To explore the safety and efficacy of neoadjuvant therapy for locally advanced rectal cancer with short course radiotherapy followed by camrelizumab combined with fluzoparib and chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provided written informed consent form for participation in this study;
2. Aged 18-75 years old, male or female;
3. Histologically confirmed pathological diagnosis of proficient mismatch repair/microsatellite stable(pMMR/MSS) rectal adenocarcinoma;
4. The lower margin of the tumor is ≤10cm from the anal verge;
5. Clinical Stage (according to the 8th edition of AJCC) T3NanyM0 and confirmed on imaging to fulfil at least any of the following: （1）MRF (+)，（2）EMVI（+），（3）LPLN（+）；or T4NanyM0 with or without one of the above three;
6. Those who are expected to achieve R0 resection;
7. Able to swallow tablets normally;
8. Patients with the ECOG performance status of 0 or 1 at the time of enrollment;
9. Patients have not received any previous anti-tumor therapy for rectal cancer;
10. Planning to undergo surgery after completion of neoadjuvant therapy;
11. Have no contraindications to surgery;
12. Normal function of major organs, including:

    1. Routine blood tests (no blood components, cell growth factors, leukocyte boosters, platelet boosters, or anaemia-correcting drugs will be allowed within 14 days prior to the first dose of study drug):White blood cell count ≥ 4.0 x 109/L; Neutrophil count ≥ 1.5 x 109/L; Platelet count ≥100×109/L; Hemoglobin ≥90 g/L
    2. Blood biochemistry: Total bilirubin ≤ 1.5 x ULN; ALT ≤ 2.5×ULN, AST ≤ 2.5×ULN; Serum creatinine ≤ 1.5 x ULN, or creatinine clearance ≥ 50 mL/min (Cocheroft-Gault formula)
    3. Coagulation: International normalised ratio (INR) ≤ 1.5 x ULN; Activated partial thromboplastin time (APTT) ≤ 1.5×ULN
13. Female subjects of childbearing potential are required to have a negative serum pregnancy test within 72 hours prior to initiation of study drug administration and to use effective contraception (e.g., intrauterine device, birth control pills, or condoms) during the trial period and for at least 3 months after the last dose of study drug; for male subjects whose partner is a female of childbearing potential, effective contraception should be used during the trial period and for 3 months after the last dose of study drug; and for male subjects whose partner is a female of childbearing potential, effective contraception should be used during the trial period and for 3 months after the last dose of study drug. Use effective contraception;

Exclusion Criteria:

1. A pre-existing history of allergy to monoclonal antibodies, any component of camrelizumab, fluzoparib, capecitabine, oxaliplatin, or other platinum-based drugs;
2. Has received, or is receiving, any of the following prior treatments：a) Any radiotherapy, chemotherapy, or other antineoplastic drug directed against the tumor; b) Treatment with immunosuppressive drugs, or systemic hormonal drugs for immunosuppression (doses > 10 mg/day prednisone or equivalent) within 2 weeks prior to first use of study drug; inhaled or topical steroids and adrenocorticotropic hormone replacement at doses > 10 mg/day prednisone or equivalent are permissible in the absence of active autoimmune disease; c) Received a live attenuated vaccine within 4 weeks prior to first use of study drug; d) Major surgery or severe trauma within 4 weeks prior to first use of study drug;
3. Any active autoimmune disease or history of autoimmune disease including, but not limited to: interstitial pneumonitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered for inclusion after hormone replacement therapy); patients with psoriasis or childhood asthma/allergies that have been in complete remission and do not require any intervention in adulthood may be considered for inclusion, but patients requiring bronchial Medical intervention with bronchodilators may not be included;
4. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation or allogeneic bone marrow transplantation;
5. Presence of cardiac clinical conditions or diseases that are not well controlled, including, but not limited to, such as (1) NYHA Class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmia that is not clinically intervened with or that remains poorly controlled after clinical intervention;
6. A serious infection (CTCAE > grade 2) within 4 weeks prior to first use of study drug, such as severe pneumonia, bacteremia, or infectious co-morbidities requiring hospitalisation; except for prophylactic antibiotics if baseline chest imaging suggests active lung inflammation, signs and symptoms of infection within 14 days prior to first use of study drug, or if oral or intravenous antibiotic therapy is required ;
7. The presence of active tuberculosis infection by history or CT scan, or a history of active tuberculosis infection within 1 year prior to enrolment, or a history of active tuberculosis infection more than 1 year ago without regular treatment
8. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV RNA above the lower detection limit of the analytical method);
9. Other malignancies diagnosed within 5 years prior to the first use of study drug, unless malignancies with a low risk of metastasis or risk of death (5-year survival >90%), such as adequately treated basal cell carcinoma of the skin or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix, may be considered for enrolment;
10. Women during pregnancy or lactation;
11. In the judgement of the investigator, the presence of other factors that may lead to forced termination of the study in the middle of the study, such as the presence of other serious illnesses (including psychiatric illnesses) that require comorbid treatment, alcoholism, drug abuse, family or social factors that may affect the safety of or compliance with the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 36 months
  Incidence and grade according to NCI-CTCAE 5.0(including serious adverse events and immune-related adverse events); Surgical safety: surgical complications, 30 - and 90-day postoperative mortality, length of stay, and reoperation rate
pCR (Pathological Complete Response) | up to 6 months
  The proportion of subjects with no residual viable tumor cells(ypT0N0) in the primary tumor and lymph nodes, also defined as the proportion of subjects with grade 0 in the AJCC Tumor Regression Grading (TRG) scoring system(version 8.0).

SECONDARY OUTCOMES:
3-year Event-Free Survival(EFS) rate | up to 36 months
  The percentage of patients without disease recurrence or progression or death due to any cause after 3-year follow-up
Overall Survival(OS) | up to 36 months
  The time from the date of randomization to the death caused by any cause
R0 resection rate | up to 6 months
  The rate of negative margin microscopically
Completion rate of neoadjuvant therapy | up to 6 months
  the rate of NAT completion
Tumor Regression grade (TRG) | up to 6 months
  Evaluated according to AJCC Version 8 TRG scoring system
quality of life (QOL) | up to 36 months
  The EORTC QLQ-C30 scale was used

OTHER OUTCOMES:
biomark | up to 36 months
  evaluate the relationship between potential biomarkers (including but not limited to MMR status, PD-L1 expression) and efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China